CLINICAL TRIAL: NCT03739489
Title: Effects of Repetitive Transcranial Magnetic Stimulation on Heart Rate Variability
Acronym: TMSXHRV
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Ricardo Galhardoni, assistant professor, Clinical Research, University of Sao Paulo
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: RG-02
Record Dates: First submitted 2018-03-28; First posted 2018-11-13 (Actual); Last update posted 2018-11-13 (Actual); Status verified 2018-11

CONDITIONS: Heart Rate Variability
Keywords: healthy subjects; repetitive transcranial magnetic stimulation; heart rate variability
MeSH Terms: interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: The participant will be received three different sessions of rtms, with wash out 30 days between sessions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- rTMS-PSI (Active Comparator): Participants allocated in this arm will receive active repetitive transcranial magnetic stimulation over the posterior superior insula right.
  Interventions: Procedure: Repetitive transcranial magnetic stimulation
- rTMS-M1 (Active Comparator): Participants allocated in this arm will receive active repetitive transcranial magnetic stimulation over the right primary motor cortex.
  Interventions: Procedure: Repetitive transcranial magnetic stimulation
- rTMS-F3 (Active Comparator): Participants allocated in this arm will receive active repetitive transcranial magnetic stimulation over the left pre frontal dorsolateral cortex.
  Interventions: Procedure: Repetitive transcranial magnetic stimulation

INTERVENTIONS:
Procedure: Repetitive transcranial magnetic stimulation — Repetitive transcranial magnetic stimulation was a technique able to modulate the brain circuit restoring the function.

SUMMARY:
Repetitive transcranial magnetic stimulation is a non-invasive neuromodulation technique used to treat different neuropsychiatric disorders, such as, depression, neuropathic pain, fibromyalgia and obsessive-compulsive disorder. It is known that the heart rate variability is altered in these conditions. Therefore the focus of this research is to show the influence of rTMS on the Heart Rate Variability.

ELIGIBILITY:
Inclusion Criteria:

* Agreed participate the protocol
* Signing the consent form
* Do not present any cardiac problems or disease

Exclusion Criteria:

* Trauma of Skull, epilepsy don't treated,
* Use of medications decrease the seizure threshold
* Patients in use of drugs, how cocaine and alcohol
* Neurosurgical clips, pacemakers, increased intracranial pressure (risk of sequelae after seizure)
* Pregnant or breastfeeding women

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-04-01 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Heart rate variability changes | Three times during the entire study. Following the scheme, Until 1 hour before each session, 15 minutes along the each session and until 1 hour after the end of session
  Changes in heart rate variability measured by Polar V800

SECONDARY OUTCOMES:
Conditioned Pain Modulation | 48 hours before the first session of stimulation
  change in pain units on a scale of 0-100. 0 no pain. 100 = the maximum pain
Volume in | 1 week before the first session of stimulation
  Determine if volume cortical regions can serve as biomarkers to predict rTMS treatment response in Healthy volunteers

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo (HC/FMUSP), São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No